CLINICAL TRIAL: NCT05370105
Title: Characterization of Circulating Extracellular Vesicles/Exosomes as New Predictive Biomarkers in Stroke Patients
Brief Title: Extracellular Vesicles as Stroke Biomarkers
Acronym: EXO4STROKE
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Other Study IDs: EXO4STROKE
Record Dates: First submitted 2022-03-22; First posted 2022-05-11 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Stroke; Rehabilitation
Keywords: brain remodeling; extracellular vesicles; biosensor; biophotonics; rehabilitation markers; regeneration; neuroinflammation; stroke biomarkers
MeSH Terms: conditions — Stroke; Neuroinflammatory Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples used for extracellular vesicles isolation. DNA content will be not considered
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke patients: 80 post-stroke patients will be asked to undergo three samples of biological material (10 ml of blood): the first collection on the second day of hospitalization at IRCCS S. Maria Nascente (Milano) or at IRCCS Don Gnocchi (Florence) of Fondazioen Don Gnocchi (t0) and a second withdrawal at discharge (t1), or approximately 2 months after the first withdrawal. Where possible, a third sampling (t2 - follow up) will be performed 6 months after the event.
  Interventions: Other: blood withdrawal
- Healthy Controls: The healthy controls will be volunteers recruited at Fondazione Don Gnocchi, who are not affected by neurodegenerative and cardiovascular diseases and who have not taken anti-inflammatory drugs in the week prior to recruitment.
  Interventions: Other: blood withdrawal

INTERVENTIONS:
Other: blood withdrawal — 10 ml of blood, two 5 ml tubes suitable for serum isolation. Given the nature and objectives of the study, there are no risks and / o inconveniences of particular importance for the patient since the blood samples will be performed according to the common procedure used in all analysis laboratories. At the end of the collection, in the area where the blood sample was taken, a small bruise may form which will disappear in the following hours, in any case during the collection particular attention will be paid to the subjects being treated with antiplatelet and anticoagulants.
  The study does not include the execution of interventional treatments or therapies.

SUMMARY:
The combination of rehabilitation protocols and regenerative therapies offers the outstanding opportunity to promote and enhance the endogenous regenerative and repair processes occurring in tissues damaged or lost due to injury, disease, or age. Still, one of the main hurdles in the clinical approach to regenerative rehabilitation is the lack of easily accessible and sensitive biomarkers for the evaluation of rehabilitation and therapy efficacy. Extracellular vesicles (EVs) are nanoscaled vesicles that mediate intercellular communication among organs. EVs were shown to be involved in the onset, progression and resolution of many disorders, being also used as valuable tool in the regenerative medicine field. However, the initial enthusiastic approach to EVs has been hindered in its transfer to clinics because of technological obstacles related to their dimensions and to their limited amount. The present project proposes the application of a Surface Plasmon Resonance imaging (SPRi)-based biosensor for the detection and characterization of blood EVs from stroke patients, before and after rehabilitation. After the successful SPRi detection of EVs of different cellular origin (brain and non-brain cells), the quantification of specific surface molecules related to pathological or regeneration processes will be accomplished. If successful, the project will 1) demonstrate the ability of the SPRi biosensor to reveal differences in the relative amount of specific cell-derived EV subpopulations and in their cargo during disease progression and rehabilitation induced recovery, 2) provide support for using the proposed SPRi-based biosensor for the detection and characterization of circulating EVs in order to evaluate the efficacy of rehabilitation protocols and regenerative therapies, 3) identify new biomarkers for the profiling of stroke patients to personalize the rehabilitation therapies.

DETAILED DESCRIPTION:
OBJECTIVE: The aim of the project will be the evaluation of the prognostic power of circulating extracellular vesicles (EVs) in the serum of stroke patients. The characterization by SPRi of different families of EVs will allow to evaluate the activation status of the processes of neuroinflammation, neuronal regeneration, angiogenesis and cellular damage to provide a picture of the mechanisms of response to the damage taking place in the patient. These data will be correlated with emerging prognostic markers derived from the literature (Gandolfi et al, 2017) and with the outcome of the rehabilitation evaluated with specific functional and neurological scales that allow accurate profiling of the patient and the evaluation of functional recovery, according to what recently validated in the "Minimum rehabilitation evaluation protocol of the person with Cerebral Stroke Version 2020 - PMIC 2020" by the Italian Society of Physical and Rehabilitative Medicine (SIMFER) (https://springerhealthcare.it/mr/numero/volume-34-n- 2-June-2020 /).

The PMIC 2020 aims to provide each physiatrist / Rehabilitation Team with a uniform tool for the assessment of the person with stroke in the different phases of the disease, from acute hospital to territorial rehabilitation.

Specific objectives will be:

i) optimization of the SPRi method for the identification of different families of EVs in the serum of healthy subjects; ii) evaluation of the feasibility of the SPRi based method for the characterization of EVs from the serum of stroke patients; iii) preliminary study of the correlation between SPRi data, soluble markers of inflammation and regeneration, patient profiling and rehabilitation outcome at discharge.

IMPACT: The personalization of the rehabilitation plan in relation to the injury suffered and the patient's active response would lead to an increased probability of functional recovery, with benefits in terms of quality of life for the patient and family members, and a reduction in the management costs of the for the National Health System.

SAMPLE COLLECTION: 80 post-stroke patients will be asked to undergo three samples of biological material (10 ml of blood, two 5 ml tubes suitable for serum isolation): the first collection on the second day of hospitalization (t0) at IRCCS S. Maria Nascente (Mialno) or IRCCS Don Gnocchi (Florence) of Fondazioen Don Gnocchi; a second withdrawal at discharge (t1), or approximately 2 months after the first withdrawal. Where possible, a third sampling (t2 - follow up) will be performed 6 months after the event at the IRCCS S. Maria Nascente or at the IRCCS in Florence. 20 healthy subjects will be asked to undergo a single sample of biological material (10 ml of blood, two 5 ml tubes suitable for serum isolation).

EV ISOLATION: The blood sample will be processed for serum separation. The samples will be coded, sterile aliquoted and stored at -80°C at the Laboratory of Nanomedicine and Clinical Biophotonics of IRCCS S. Maria Nascente (Milan) until used.

EVs will be isolated from serum by size exclusion chromatography (qEV; Izon). The actual isolation will be verified with standard techniques, including for example western blot for specific protein markers (CD63, Flotillin 1), Nanoparticle Tracking Analysis or Transmission Electron Microscopy.

SPRi BIOSENSOR: The functionalization of the SPRi chip will be optimized for known markers of apoptotic bodies (Annexin V; index of extent of brain damage) and of EVs from neurons (Ephrin), microglia (IB4 or CD11b), astrocytes (GLAST) and endothelial cells ( CD31). The chip will be also functionalized for the recognition of the Klotho protein (Sahu et al, 2018).

Immobilized EVs will be tested also for the presence on the surface of receptors related to neuronal regeneration (TGFbR1 / 2), microglial activation (TSPO) and angiogenesis (VEGFR-2).

RAMAN ANALYSIS: EVs isolated from patient serum will also be analyzed by Raman spectroscopy according to a protocol already optimized for patients with Parkinson's disease(Gualerzi et al., 2019). Raman analysis will provide information on the biochemical characteristics of the EVs, which can be correlated with the molecular data obtained in SPRi.

ELISA: known markers of inflammation and neuronal activation will be quantified in serum by ELISA assays: inflammatory cytokines (IL6 and TNFa), adipokines (leptin), soluble adhesion molecules (sICAM, sFAS) and growth factors (BDNF).

Correlation between SPRi data, soluble inflammatory and neurotrophic factors will be performed to identify new rehabilitation markers for stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ischemic or haemorrhagic stroke related to intensive post-stroke rehabilitation hospitalization
* within 15 days of the ictal event

Exclusion Criteria:

* Previous head injuries/traumas
* Oncological diseases
* Diseases of the immune and haematological system
* Neurodegenerative diseases

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at Fondazione Don Gnocchi after stroke injury and undergoing an intensive rehabilitation program.
Sampling Method: Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in modified Barthel index after rehabilitation | 01/11/2020 - 30/03/2022
  modified Barthel index (Shah et al., 1989)

SECONDARY OUTCOMES:
Extracellular vesicles characterization by SPRi | 25/06/2018 - 30/09/2022
  EVs will be isolated from serum, characterized by standard procedures and injected on the SPRi biosensor for the differential quantification of multiple EV subfamilies. Secondary antigens will be evaluated on the surface of immobilized EVs.
  Changes in biomarkers expression will be assessed after rehabilitation
Change in Numeric Rating Scale (NRS) PAIN or PAINAD for non-verbal patient after rehabilitation | 25/06/2018 - 30/09/2022
  Numeric Rating Scale (NRS) PAIN or PAINAD for non-verbal patient, validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in anamnestic and current modified RANKIN scale after rehabilitation | 25/06/2018 - 30/09/2022
  anamnestic and current modified RANKIN scale, validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in NIH-STROKE SCALE after rehabilitation | 25/06/2018 - 30/09/2022
  NIHSS scale (Brott et al. 1989) , validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in Fugl-Meyer Assessment (FMA) scale after rehabilitation | 25/06/2018 - 30/09/2022
  Fugl-Meyer Assessment (FMA) scale (Fugl-Meyer et al., 1975; Cecchi et al., 2020) , validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in Trunk control test after rehabilitation | 25/06/2018 - 30/09/2022
  Trunk control test (Franchignoni et al, 1997), validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in Short Physical Performance Battery (SPPB) after rehabilitation | 25/06/2018 - 30/09/2022
  SPPB (Guralnik et al, 1994) , validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in Functional ambulation classification | 25/06/2018 - 30/09/2022
  Functional ambulation classification (Jan Mehrholz et al., 2007), validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in Addenbrooke's Cognitive Examination scale after rehabilitation | 25/06/2018 - 30/09/2022
  Addenbrooke's Cognitive Examination (Mathuranath et al., 2000), validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in Hospital Anxiety and Depression Scale (HADS) after rehabilitation | 25/06/2018 - 30/09/2022
  HADS, validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.
Change in Cumulative illness rating scale (CIRS) after rehabilitation | 25/06/2018 - 30/09/2022
  CIRS (Linn et al., 1968), validated in the literature and already proposed in the PMIC 2020 by SIMFER, will be used for accurate patient profiling and assessment of functional recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Gualerzi, PhD, Principal Investigator — Fondazione Don Carlo Gnocchi, Laboratory of Nanomedicine and Clinical Biophotonics
Locations (2):
- Italy (2):
  - IRCCS Don Gnocchi, Fondazione Don Carlo Gnocchi ONLUS, Florence
  - IRCCS S. Maria Nascente, Fondazione Don Carlo Gnocchi ONLUS, Milan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Picciolini S, Gualerzi A, Vanna R, Sguassero A, Gramatica F, Bedoni M, Masserini M, Morasso C. Detection and Characterization of Different Brain-Derived Subpopulations of Plasma Exosomes by Surface Plasmon Resonance Imaging. Anal Chem. 2018 Aug 7;90(15):8873-8880. doi: 10.1021/acs.analchem.8b00941. Epub 2018 Jul 17. PMID 29972017
- [Background] Gualerzi A, Picciolini S, Carlomagno C, Terenzi F, Ramat S, Sorbi S, Bedoni M. Raman profiling of circulating extracellular vesicles for the stratification of Parkinson's patients. Nanomedicine. 2019 Nov;22:102097. doi: 10.1016/j.nano.2019.102097. Epub 2019 Oct 21. PMID 31648040
- [Background] Picciolini S, Gualerzi A, Carlomagno C, Cabinio M, Sorrentino S, Baglio F, Bedoni M. An SPRi-based biosensor pilot study: Analysis of multiple circulating extracellular vesicles and hippocampal volume in Alzheimer's disease. J Pharm Biomed Anal. 2021 Jan 5;192:113649. doi: 10.1016/j.jpba.2020.113649. Epub 2020 Sep 23. PMID 33038641
- [Background] Gualerzi A, Picciolini S, Carlomagno C, Roda F, Bedoni M. Biophotonics for diagnostic detection of extracellular vesicles. Adv Drug Deliv Rev. 2021 Jul;174:229-249. doi: 10.1016/j.addr.2021.04.014. Epub 2021 Apr 19. PMID 33887403
- [Background] Gualerzi A, Picciolini S, Roda F, Bedoni M. Extracellular Vesicles in Regeneration and Rehabilitation Recovery after Stroke. Biology (Basel). 2021 Aug 30;10(9):843. doi: 10.3390/biology10090843. PMID 34571720
- [Result] Picciolini S, Mangolini V, Roda F, Montesano A, Arnaboldi F, Liuzzi P, Mannini A, Bedoni M, Gualerzi A. Multiplexing Biosensor for the Detection of Extracellular Vesicles as Biomarkers of Tissue Damage and Recovery after Ischemic Stroke. Int J Mol Sci. 2023 Apr 27;24(9):7937. doi: 10.3390/ijms24097937. PMID 37175644
- See also: Laboratory of Nanomedicine and Clinical Biophotonics, Fondazione Don Carlo Gnocchi — http://www.labion.eu